CLINICAL TRIAL: NCT06785922
Title: Differences in Gastric Microbiota in Patients Who Were Infected Between CagA Positive and Negative Helicobacter Pylori
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Si 224/2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Gastric Microbiota; Helicobacter Pylori; CagA; Gastric Cancer
Keywords: Gastric microbiota; Helicobacter pylori; CagA; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CagA positive H.pylori (Other): CagA positive H.pylori
  Interventions: Procedure: Stomach biopsy for gastric microbiota
- CagA negative H.pylori (Other)
  Interventions: Procedure: Stomach biopsy for gastric microbiota

INTERVENTIONS:
Procedure: Stomach biopsy for gastric microbiota — Stomach biopsy for gastric microbiota testing (16S RNA sequencing)

SUMMARY:
The goal of this clinical trial is to study the differences in gastric microbiota (Diversity index) between patients who were infected with CagA-positive Helicobacter pylori and CagA-negative Helicobacter pylori. The main question it aims to answer are:

The effect of Helicobacter pylori typing (CagA status) on gastric microbiota, what is the different?

Patients indicated for EGD at Siriraj Endoscopic Center will undergo a Helicobacter pylori test (Rapid urease test) If the result is positive, a stomach biopsy for gastric microbiota testing and CagA antibody testing will be conducted. Then, the patients will be divided into two groups: CagA-positive Helicobacter pylori and CagA-negative Helicobacter pylori.

To compare the differences in gastric microbiota in terms of species and biodiversity, as well as endoscopic results, etc.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 with an indication for EGD
* Helicobacter pylori infection (Rapid urease test positive)

Exclusion Criteria:

* Severe comorbidities: poorly controlled DM, ESRD, decompensated cirrhosis, Malignancy
* BMI ≤ 23 kg/m2
* Receiving medications that affect the gastric microbiota include Antibiotics, probiotics, or bismuth within 4 weeks, PPI within 2 weeks, NSAIDs or Metformin within 2 weeks
* History of cholecystectomy or proximal small bowel surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The differences in gastric microbiota (Diversity index) | On the 1 day of EGD
  Diversity index: Shannon index, Simpson index

SECONDARY OUTCOMES:
Microbiota composition | On the 1 day of EGD
  Prevalence of microbiota species
Endoscopic finding | During the EGD
  Endoscopic finding was described by investigators
Pathological finding | Within 2 week after EGD
  Pathological finding was described by pathologist

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of internal medicine siriraj hospital, Mahidol university, Bangkok Noi, Bangkok, Thailand